CLINICAL TRIAL: NCT03624374
Title: Characterization of the Natural History of Leukoencephalopathy With Brainstem and Spinal Cord Involvement and Lactate Elevation
Brief Title: Natural History Study of Leukoencephalopathy With Brainstem and Spinal Cord Involvement and Lactate Elevation (LBSL)
Status: Recruiting | Type: Observational
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00150619
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Leukoencephalopathies; LBSL; Leukoencephalopathy With Brainstem and Spinal Cord Involvement and Lactate Elevation; White Matter Disease; Ataxia, Cerebellar; Genetic Disease
Keywords: Natural History Study; Kennedy Krieger Institute; Virtual assessment; DARS2; Johns Hopkins Hospital
MeSH Terms: conditions — Leukoencephalopathies; Leukoencephalopathy with Brainstem and Spinal Cord Involvement and Lactate Elevation; Cerebellar Ataxia; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we will conduct retrospective chart and imaging reviews and prospective longitudinal virtual assessments of individuals with LBSL.

DETAILED DESCRIPTION:
LBSL (leukoencephalopathy with brainstem and spinal cord involvement and lactate elevation) is a rare genetic disorder characterized by slowly progressive cerebellar ataxia and spasticity with dorsal column dysfunction (decreased position and vibration sense) in most patients. Manual dexterity becomes impaired to a variable degree. Associated problems include dysarthria, mild cognitive decline and learning problems, and epilepsy. LBSL is diagnosed by identification of biallelic pathogenic variants in DARS2, encoding mitochondrial aspartyl tRNA synthetase and characteristic abnormalities observed on the brain and spinal cord MRI. Most of the literature consists of case reports and case series and there are only limited data that provide details on genotype-phenotype correlations. There is very little quantitative or semi-quantitative information about neurocognitive and neuromotor impairment in LBSL. There are currently no targeted therapies or guidelines about supportive therapies for LBSL.

In this study, we will conduct retrospective chart and imaging reviews and prospective longitudinal virtual assessments of individuals with LBSL.

We hypothesize that 1) there will be a broad phenotypic spectrum of neuromotor and neurocognitive deficits in LBSL patients; 2) most impairment will likely be related to gait; 3) there will be a threshold of impairment in gait that is associated with poorer quality of life for these patients; 4) and that even in patients with apparently mild disease there will be neurocognitive deficits related to cortical and cerebellar white matter abnormalities.

Answering these hypotheses will form the basis of a better understanding of the natural history of LBSL. It will help further characterize the expected level of impairment based on a patient's genotype. This will be particularly helpful for providing anticipatory guidance for newly diagnosed infants and children with LBSL. The information will also help identify priorities for existing supportive therapies and help clarify the common or clinically meaningful symptoms that should be targeted for new treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed DARS2 mutation through genetic analysis
2. Ability of the caregiver or participant to speak and understand English at an 8th-grade level

Exclusion Criteria:

* The vulnerable populations of prisoners, non-viable neonates, pregnant women, adults lacking the capacity to consent, non-English speakers or children who are in foster care or wards of the state.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All case subjects will be known to have leukoencephalopathy with brainstem and spinal cord involvement and lactate elevation.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Track Natural History of LBSL patients using medical record review | 4/1/2018 - 3/31/2023
  Participants will be asked to provide all prior neurological, developmental and genetics medical records and available neuroimaging studies. We will first confirm eligibility by review of MRI and DARS2 mutation analysis. We will determine information about disease duration, rate of symptom progression and prevalence of specific neurological symptoms and the level of disability.
  We have derived an MRI severity score by modifying a standard leukodystrophy MRI scoring system, referred to as the Loes severity score (developed by Dr. Daniel Loes). This score is routinely used by radiologists. We will be reviewing and scoring participant neuroimages to better understand correlation with disease severity and progression.
Assessment of behavior in patients with LBSL using standardized neurocognitive surveys. | 4/1/2018 - 3/31/2023
  After the participant is enrolled, they will receive several neurocognitive assessments that will be sent digitally, including the Child or Adult Behavior Checklist (CBCL/ABCL). The CBCL/ABCL is one of most widely used measures in psychology to identify behavioral problems or mood disorders in children or adults, respectively. The scoring of this checklist is grouped by eight empirically based syndrome scales. These include aggressive behavior, anxious/depressed, attention problems, rule-breaking behavior, somatic complaints, social problems, thought problems, withdrawal/depression symptoms. The CBCL has standardized scores for children of the same gender and similar age and are interpreted as falling in the normal, borderline, or clinical range.
Assessment of social communication in patients with LBSL using standardized neurocognitive surveys. | 4/1/2018 - 3/31/2023
  After the participant is enrolled, they will receive several neurocognitive assessments that will be sent digitally, including the Social Communication Questionnaire (SCQ) The SCQ used by the International Autism Network will be used to screen individuals for Autism Spectrum Disorder and is completed by a caregiver. The SCQ is a 40 item, parent report screening measure that identifies whether a child has the associated symptoms of autism spectrum disorder.
Assessment of executive function in patients with LBSL using standardized neurocognitive surveys. | 4/1/2018 - 3/31/2023
  After the participant is enrolled, they will receive several neurocognitive assessments that will be sent digitally, including the Behavioral Rating Inventory of Executive Function (BRIEF).The BRIEF assesses impairment of executive function by evaluating eight clinical scales of executive function including inhibit, shift, emotional control, initiate, working memory, plan/organize, organization of materials, and monitor.The BRIEF exists for preschool children (2-5) and there are self-report versions for adolescents and adults.
Assessment of adaptive function in patients with LBSL using standardized neurocognitive surveys. | 4/1/2018 - 3/31/2023
  After the participant is enrolled, they will receive several neurocognitive assessments that will be sent digitally, including the Adaptive Behavior Assessment System version 3 (ABAS-3). The ABAS-3 survey assesses eleven essential skill areas in 3 major adaptive domains including conceptual, social and practical, and assists in diagnosing various developmental, learning, and behavioral disabilities. This complete battery of adaptive skills can be administered across the life span for ages Birth-89 years.
Assessment of quality of life in patients with LBSL using standardized surveys. | 4/1/2018 - 3/31/2023
  After the participant is enrolled, they will receive several quality of life assessments that will be sent digitally. Information on quality of life in LBSL will be collected using well-validated scales addressing physical, emotional, social and school functioning. Relevant scales include quality of life in children and adults with spasticity, quality of life in children and adults with ataxia, and quality of life in children and adults with chronic medical conditions.
Assessment of ataxia in patients with LBSL using wearable sensor technology and standardized clinical scales. | 4/1/2018 - 3/31/2023
  The study team will collect information about ataxia using wearable sensors and by administering the Standardized Assessment and Rating of Ataxia (SARA) scale at participant's homes.
  The SARA scale is an 8-item performance based scale that assesses upper and lower extremity ataxia. A total score of 0 indicates no ataxia and the maximum score of 40 indicates severe ataxia.
Assessment of balance in patients with LBSL using wearable sensor technology. | 4/1/2018 - 3/31/2023
  The study team will collect information about gait and balance ability over time using functional surveys as well as wearable sensors to be used at the participant's homes.
  This series of tests will require the participant to stand in several different poses for 2 trials of 30 seconds each to assess their balance. This will include standing with their eyes open and their feet apart and together, as well as with their eyes closed and their feet apart and together.
Timed Up and Go Test | 4/1/2018 - 3/31/2023
  This test will require the participant to sit in a chair. When the participant is instructed to, they will stand up from the chair, walk 3 meters in a straight line, turn around and walk back to the chair. The test duration and variables such as walking and turning speed will be obtained.
Long Walk Test | 4/1/2018 - 3/31/2023
  This test will require the participant to walk 22 feet in a straight line for a duration of 2 minutes. Variables such as walking and turning speed, stride length and step-to-step variability will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Amena S Fine, MD PhD, Principal Investigator — Moser Center for Leukodystrophies at Kennedy Krieger Institute
Locations (1):
- Hugo Moser Center for Leukodystrophies, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No